CLINICAL TRIAL: NCT03044600
Title: Gene Expression in Hyperparathyroidism: Identifying Molecular Differences in MEN1 Patients Versus Young MEN1 Negative Patients
Brief Title: Gene Expression in Hyperparathyroidism
Status: Terminated | Type: Observational
Why Stopped: At the request of the Principal Investigator
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA12-0944
Record Dates: First submitted 2017-02-03; First posted 2017-02-07 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Parathyroid Disease; Hyperparathyroidism
Keywords: Parathyroid disease; Hyperparathyroidism; Chart review; MEN1-negative; HRPT2 mutations
MeSH Terms: conditions — Parathyroid Diseases; Hyperparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Parathyroid tissue previously obtained during surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young MEN1 Negative Group: Participants under 50 years of age who have been diagnosed with MEN1-negative primary hyperparathyroidism.
  Interventions: Other: Chart Review; Other: HRPT2 Mutation Evaluation

INTERVENTIONS:
Other: Chart Review — Patient charts will be reviewed to collect demographic data, pre-operative and post-operative clinical and laboratory data, operative reports, and pathology reports.
Other: HRPT2 Mutation Evaluation — Archived formalin-fixed paraffin-embedded (FFPE) tissue blocks from surgical specimens of patients stained for parafibromin to evaluate for HRPT2 mutations.

SUMMARY:
Objectives:

1. To better define the differences in molecular genetics of parathyroid tumors in patients with MEN1, single gland parathyroid disease in patients less than 50 years old and single gland disease in patients greater than 50 years old.
2. To better define the incidence of HRPT2 mutation in young patients with primary hyperparathyroidism and determine whether routine testing in these patients is indicated.

DETAILED DESCRIPTION:
Patient charts will be reviewed to collect demographic data, pre-operative and post-operative clinical and laboratory data, operative reports, and pathology reports. Archived formalin-fixed paraffin-embedded (FFPE) tissue blocks from surgical specimens of patients will be stained for parafibromin to evaluate for HRPT2 mutations.

ELIGIBILITY:
Inclusion Criteria:

1. All patients previously enrolled in parathyroid tissue banking under protocol Lab08-0034.
2. For the subgroup designated for HRPT2 mutation testing:

Patients with primary hyperparathyroidism who are younger than 50 years of age and have tested negative for MEN1, between January 1, 1980 and the present.

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with parathyroid tumors at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-10-18 (Actual)

PRIMARY OUTCOMES:
Molecular Genetics of Parathyroid Tumors | 10 years
  RNA isolated from banked frozen tissues. cDNA microarray prepared using an Illumina array chip. Results analyzed using Ingenuity analysis software to detect 2-fold changes in gene expression. T-statistics used to determine significantly discriminating genes.

SECONDARY OUTCOMES:
HRPT2 Mutations | 10 years
  Archived formalin-fixed paraffin-embedded (FFPE) tissue blocks from surgical specimens of patients stained for parafibromin to evaluate for HRPT2 mutations.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy D. Perrier, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org